CLINICAL TRIAL: NCT06971939
Title: A Phase 4, Multicenter, Open-label Study to Evaluate Long-term Safety and Efficacy of Revakinagene Taroretcel-Lwey (NT-501) Previously Implanted During a Phase 1, Phase 2, or Phase 3 Clinical Study and to Evaluate NT-501 Implanted in Participants Who Underwent the Sham Procedure in a Phase 3 Clinical Study of Macular Telangiectasia Type 2 (MacTel)
Brief Title: Phase 4 Study: Long-term Safety and Efficacy of NT-501 in MacTel Type 2, Including Sham Procedure Participants
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTMT-04
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Macular Telangiectasia Type 2 (MacTel)
Keywords: Ciliary Neurotrophic Factor (CNTF); Macular Telangiectasia Type 2 (MacTel)

STUDY DESIGN:
Intervention Model Description: Arms 1 and 2: For participants who previously received a single NT-501, the implanted eye is designated the study eye. For participants who received an NT-501 implant in both eyes (ie. the first implant received in NTMT-01, NTMT-02, NTMT 01/02E, NTMT-03-A, or NTMT-03-B, and the second implant received in NTMT-02B), both eyes will be designated as study eyes (the eye in which NT-501 was originally implanted will be study eye 1 and the other implanted eye will be study eye 2).
  Arm 3: The implanted eye will be designated as the study eye in Arm 3. Note, if NT-501 in not implanted in the Sham eye (ie. the eye that did not undergo intervention during the parent Phase 3 clinical study), then the sham eye will also be considered a study eye for long-term follow-up.
  Regardless of study eye designation, both eyes of each participant in all 3 study arms will be evaluated during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Arm 1 (Phase 3 Long-term Follow-up) (Other): For participants who received NT-501 (ENCELTO) in a previous Phase 3 study (NTMT-03-A or NTMT-03-B), or for participants who received NT-501 (ENCELTO) in both eyes (i.e. participated in study NTMT-02B) but received the first NT-501 (ENCELTO) implant in a Phase 3 study. No new treatment intervention will be administered. Arm 2 is focused on long term follow-up for participant who already has the ENCELTO implant at time of study screening and enrollment.
  Interventions: Combination Product: NT-501/revakinagene taroretcel-lwey
- Arm 2 (Phase 1 and Phase 2 Long-term Follow-up) (Other): For participants who received NT-501 (ENCELTO) in a previous Phase 1 study (NTMT-01), Phase 2 study (NTMT-02), in the sub study of Phase 1 and Phase 2 extension study (NTMT-01/02E), or for participants who received NT-501 (ENCELTO) in both eyes (i.e. participated in study NTMT-02B) but received the first NT-501 (ENCELTO) implant in a Phase 1 or Phase 2 study. No new treatment intervention will be administered. Arm 2 is focused on long term follow-up for participant who already has the ENCELTO implant at time of study screening and enrollment.
  Interventions: Combination Product: NT-501/revakinagene taroretcel-lwey
- Arm 3 (Phase 3 Sham to Implant Crossover) (Experimental): For participants who underwent Sham procedure in either Phase 3 study (NTMT-03-A or NTMT-03-B) and will receive NT-501 in this study.
  Interventions: Combination Product: NT-501/revakinagene taroretcel-lwey

INTERVENTIONS:
Combination Product: NT-501/revakinagene taroretcel-lwey — NT-501 is surgically implanted into the vitreous cavity to continuously release recombinant human ciliary neurotrophic factor (CNTF).
  Other Names: ENCELTO

SUMMARY:
The purpose of this global, multicenter, open-label, Phase 4 clinical extension study is to evaluate the long-term safety and efficacy of revakinagene taroretcel-lwey (Encelto™; hereinafter referred to as NT-501), in participants with macular telangiectasia type 2 (MacTel) who previously received the intraocular implant in a Phase 1, Phase 2, or Phase 3 clinical study. In addition, this study will evaluate the safety and efficacy of NT501 in participants who previously underwent the sham procedure in a Phase 3 MacTel clinical study and elect to have NT-501 implanted intraocularly in this Phase 4 study.

DETAILED DESCRIPTION:
This extension study consists of 3 arms:

* Arm 1 (Phase 3 Treated Participants' Long-term Follow-up): Arm 1 is to assess the long-term safety and efficacy of NT-501 in participants who received NT-501 in a previous MacTel Phase 3 clinical study (NTMT-03-A or NTMT-03-B).
* Arm 2 (Phase 1 and Phase 2 Long-term Follow-up): Similar to Arm 1, Arm 2 is to assess the long-term safety of NT-501 in participants who received NT-501 in a previous MacTel Phase 1 or Phase 2 clinical study (NTMT-01, NTMT-02, or NTMT-01/02E).
* Arm 3 (Phase 3 Sham to Implant Crossover): Arm 3 will evaluate the safety and efficacy of NT-501 in participants who previously underwent the sham procedure in a Phase 3 MacTel clinical study (NTMT-03-A or NTMT-03-B) and elect to have NT-501 implanted intraocularly in this extension study.

Arms 1 and 2 are noninterventional and observational studies. Participants who received NT-501 in both eyes (ie, participated in study NTMT-02B) will be enrolled in either Arm 1 or Arm 2 based on the study in which the first NT-501 was implanted (ie, participants who received the first implant in a Phase 3 study will be enrolled in Arm 1 and those who received the first implant in the Phase 1 study or Phase 2 study will be enrolled in Arm 2).

Only Arm 3 is an interventional study where participants will receive an NT-501 implant. A participant can receive NT-501 in either eye that meets eligibility criteria according to investigator assessment, and in accordance with participant choice.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this study, an individual participant must meet all the following criteria:

1. Male or female adult participants who previously completed an NT-501 MacTel clinical study and:

   1. Arm 1: received NT-501 intraocular implant in either Phase 3 study (NTMT-03-A or NTMT-03-B)
   2. Arm 2: received NT-501 intraocular implant in the Phase 1 study (NTMT-01), Phase 2 study (NTMT-02), or in the substudy of the Phase 1 and Phase 2 extension study (NTMT-01/02E)

      Note: participants who received NT-501 in both eyes (ie, participated in study NTMT-02B) will be enrolled in either Arm 1 or Arm 2 based on the study in which the first NT 501 was implanted (ie, participants who received the first implant in a Phase 3 study will be enrolled in Arm 1 and those who received the first implant in the Phase 1 study or Phase 2 study will be enrolled in Arm 2).
   3. Arm 3: underwent the sham procedure in either Phase 3 study (NTMT-03-A or NTMT-03-B)
2. Participants must have steady fixation in the foveal or parafoveal area and sufficiently clear media for good quality retinal imaging.
3. Participant or their legally authorized representative must be able to provide written informed consent to participate in the study, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines, and local regulations, before initiating any clinical study related procedures.
4. Arm 3: female participants of childbearing potential must agree to use highly effective contraception. Highly effective forms of contraception (generally a first-year typical use pregnancy risk of 1% or less) include the following: contraceptive implants; an intrauterine device; permanent contraceptive procedures (vasectomy, bilateral salpingectomy, bilateral tubal occlusion, or partial salpingectomy); abstinence. A combination of male condom with either cap, diaphragm, or sponge with spermicide (ie, double barrier methods) is also considered an acceptable, but not highly effective, method of birth control.

Note: Participants enrolled at investigator sites in France or Germany must agree to use 2 forms of contraception listed above during study participation.

Exclusion Criteria

To participate in this study, the potential participant must not meet any of the following criteria. (Note that the ocular exclusion criteria are relevant to the study eye[s], unless indicated for both eyes):

Exclusion Criteria Applicable to Arms 1, 2, and 3:

1. Participant is medically unable to comply with clinical study procedures or visits.
2. Participant has, in the opinion of the investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations, and outcome assessments.

   Exclusion Criteria Applicable to Arm 3 Only:
3. Participant has significant corneal or media opacities in the study eye to be implanted.
4. Participant has evidence of pathologic myopia in the study eye to be implanted.
5. Participant has any of the following lens opacities in the study eye to be implanted: cortical opacity > standard 3, posterior subcapsular opacity > standard 2, or a nuclear opacity > standard 3 as measured on the Age- Related Eye Disease Study (AREDS) clinical lens grading system. Note: the participant can be reconsidered for enrollment 90 days after undergoing cataract surgery.
6. Participant has undergone lens removal in the study eye to be implanted in the previous 3 months or YAG laser within 4 weeks of the screening/baseline visit.
7. Participant has evidence of ocular disease in the study eye to be implanted other than MacTel that, in the judgment of the examining physician, may confound the diagnosis, procedures, or outcome of the study (eg. glaucoma, severe nonproliferative or proliferative diabetic retinopathy, uveitis).
8. Received intravitreal steroid therapy in the study eye to be implanted within the last year.
9. Received intravitreal anti-vascular endothelial growth factor therapy in the study eye to be implanted within the last 6 months.
10. Evidence of active exudative intraretinal neovascularization or subretinal neovascularization in the study eye to be implanted, as evidenced by hemorrhage, hard exudate, subretinal fluid, or intraretinal fluid.
11. Evidence of central serous chorioretinopathy in the study eye to be implanted.
12. Participant underwent vitrectomy, penetrating keratoplasty, trabeculectomy, or trabeculoplasty in the study eye to be implanted.
13. A history of ocular herpes virus in the study eye to be implanted.
14. Participant is on chemotherapy.
15. Participant is pregnant or breastfeeding.
16. Participation in any other clinical study of an intervention (drug or device) within 6 months prior to the screening/baseline visit.
17. A history of malignancy that would compromise survival during the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2030-08-15 (Estimated); Study Completion 2030-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular and nonocular adverse events (AEs) and serious adverse events (SAEs) | Baseline and annually for up to 5 yrs for Arms 1 and 2 and baseline, perioperative, and annually for up to 5 yrs for Arm 3 participants
  Incidence of ocular and nonocular adverse events (AEs) and serious adverse events (SAEs)
Percentage of participants with a loss of 15 letters or more in best corrected visual acuity (BCVA) compared to presurgery baseline BCVA | Baseline and annually for up to 5 yrs for Arms 1 and 2 and baseline, perioperative, and annually for up to 5 yrs for Arm 3 participants
  Percentage of participants with a loss of 15 letters or more in best corrected visual acuity (BCVA) compared to presurgery baseline BCVA using the Early Treatment Diabetic Retinopathy Study (ETDRS) distance chart

SECONDARY OUTCOMES:
Change from presurgery baseline in ellipsoid zone (EZ) area loss | Baseline and annually for up to 5 yrs for Arms 1 and 2 and baseline, perioperative, and annually for up to 5 yrs for Arm 3 participants
  Change from presurgery baseline in ellipsoid zone (EZ) area loss as measured by en face spectral domain optical coherence tomography (SD-OCT) for both eyes
Change from presurgery baseline in BCVA | Baseline and annually for up to 5 yrs for Arms 1 and 2 and baseline, perioperative, and annually for up to 5 yrs for Arm 3 participants
  Change from presurgery baseline in BCVA using the ETDRS distance chart for both eyes
Change from presurgery baseline in aggregate retinal sensitivity | Baseline and annually for up to 5 yrs for Arms 1 and 2 and baseline, perioperative, and annually for up to 5 yrs for Arm 3 participants
  Change from presurgery baseline in aggregate retinal sensitivity as measured by microperimetry within the EZ line break area for both eyes
Change from presurgery baseline in monocular reading speed | Baseline and annually for up to 5 yrs for Arms 1 and 2 and baseline, perioperative, and annually for up to 5 yrs for Arm 3 participants
  Change from presurgery baseline in monocular reading speed for both eyes
Change from presurgery baseline in the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) | Baseline and annually for up to 5 yrs for Arms 1 and 2 and baseline, perioperative, and annually for up to 5 yrs for Arm 3 participants
  Change from presurgery baseline in NEI-VFQ-25 near activities subscale score. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aaberg, Jr, MD, Study Chair — Neurotech Pharmaceuticals
Locations (33):
- United States (25):
  - Scripps Health, La Jolla, California
  - Jules Stein Eye Institute/UCLA, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Emory Eye Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Elman Retina Group, PA, Baltimore, Maryland
  - National Eye Institute, Bethesda, Maryland
  - Cumberland Valley Retina Consultants, Frederick, Maryland
  - Massachusetts Eye and Ear Infirmary, Retina Service, Boston, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Associates of Cleveland, Inc., Cleveland, Ohio
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Retina Northwest, P.C., Portland, Oregon
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Texas Retina Associates, Dallas, Texas
  - Retina Center of Texas, Dallas, Texas
  - Retina Consultants of Texas, Houston, Texas
  - University of Utah John A. Moran Center, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
- Australia (3):
  - Cerulea, East Melbourne
  - Lion's Eye Institute, Perth
  - Sydney Eye Hospital, Sydney
- Lariboisiére Hospital, Paris, France
- Germany (3):
  - University Eye Hospital Bonn, Bonn
  - UNIVERSITÄTSKLINIKUM FREIBURG, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Augenzentrum am St. Franziskus-Hospital, Münster
- Oxford University Hospitals NHS FT, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No